CLINICAL TRIAL: NCT04238923
Title: Topical Gentamicin and Vancomycin for Surgical Site Infection Prophylaxis in Patients Undergoing High-Risk Vascular Surgery
Brief Title: Topical Gentamicin and Vancomycin for Vascular Surgical Site Infection Prophylaxis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115156
Record Dates: First submitted 2020-01-22; First posted 2020-01-23 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Vascular Diseases; Peripheral Vascular Disease; Surgical Site Infection; Bypass Complication
MeSH Terms: conditions — Vascular Diseases; Peripheral Vascular Diseases; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Topical Gentamicin and Vancomycin (Experimental): Immediately prior to closure of the incision, 1g of vancomycin will be mixed in 4mL of normal saline and applied as a paste directly to the muscle, fascia and subcutaneous tissue. Gentamicin-eluting collagen sponges will be cut to the appropriate size to cover the defect and applied after application of vancomycin. Following closure, the surgical site will be covered with a sterile dressing and left in place for 48hrs.
  Interventions: Drug: Topical vancomycin paste (1g vancomycin powder + 4mL sterile saline) and Collatamp G gentamicin-eluting sponge (Azralez Pharmaceuticals; 2.0mg gentamicin sulphate/cm2 to cover wound)
- Control (No Intervention): The surgical wound is closed in the standard fashion with 3 layer closure with staples for skin. Following closure, the surgical site will be covered with a sterile dressing and left in place for 48hrs.

INTERVENTIONS:
Drug: Topical vancomycin paste (1g vancomycin powder + 4mL sterile saline) and Collatamp G gentamicin-eluting sponge (Azralez Pharmaceuticals; 2.0mg gentamicin sulphate/cm2 to cover wound) — Topical vancomycin paste and gentamicin-eluting collagen sponge will be applied directly to the deep layers of the wound following reconstruction, prior to closure.
  Arms: Topical Gentamicin and Vancomycin

SUMMARY:
Many patients who undergo vascular surgery to improve the blood flow to their legs are at risk of developing an infection in the surgical site and are then at risk of serious complications such as hospital readmission, failure of the surgical procedure and lower limb amputation. Surgical site infections may be reduced in high-risk patients by applying two commonly used antibiotics (gentamicin and vancomycin) into the surgical incision at the end of the surgical procedure. This will be compared to the standard of care treatment at London Health Sciences Center.

DETAILED DESCRIPTION:
Surgical site infections (SSI) are among the most common complications to develop following peripheral vascular surgery and increase the patient's risk for major amputation, graft failure and increase healthcare resource utilization. SSI are defined by the Center for Disease Control (CDC) as infections occurring within 30-90 days of a surgical procedure, or 1 year if a prosthetic implant was placed, and are divided into superficial, deep and organ space based on depth of microbial invasion.

The incidence of SSI in patients undergoing limb saving vascular surgery has consistently been found to exceed the CDC average of 2.1% for other clean surgical procedures, despite the routine use of perioperative antibiotics and aggressive wound care. A recent review of SSI in vascular surgery showed rates as high as 30%, and the investigators' institution has reported a SSI rate of 20%. Coagulase-negative staphylococcus species are the most frequent isolates from SSI following peripheral vascular surgery, with the highly virulent organism, MRSA becoming increasingly prevalent. Gram-negative organisms account for another 20-30% of SSI, with Pseudomonas isolates commonly identified, particularly in the groin. Several procedure- and patient-related factors have emerged as important predictors of SSI following peripheral vascular surgery, among the most important of which are obesity, tissue loss, redo surgery, dialysis dependence and diabetes mellitus. Obesity has been found to double the risk of SSI. Obese patients are shown to have lower tissue concentrations of antibiotics, which would place them at higher risk of developing SSI. Patients with tissue loss secondary to critical limb ischemia also are at increased risk of SSI resulting from bacterial spread from contaminated ulcers and poor vascular supply to the wound. As well, patients undergoing redo surgery face an increased risk of wound and graft infection secondary to the impaired vascular supply and healing potential of scar tissue. Diabetes mellitus and dialysis dependence are also independent risk factors for SSI following infrainguinal bypass due to a multitude of disease factors, especially immunologic dysfunction and impaired blood supply to the healing tissue.

Prophylactic intravenous antibiotics are the only intervention thus far consistently found to effectively prevent SSI in patients undergoing vascular surgery, however because of the aforementioned factors such measures are less effective in high-risk patients. Data to support other perioperative practices to prevent wound infections in vascular surgery are sparse. Among other surgical disciplines, topical antibiotics are re-emerging as a valid strategy to prevent SSI based on improved understanding of the mechanisms of drug delivery and identification of high-risk patients. In particular, vancomycin applied directly to surgical wounds has shown promise in preventing SSI. Topical vancomycin is believed to prevent gram-positive SSI, particularly those caused by MRSA, while minimizing adverse events related to systemic exposure to vancomycin such as nephrotoxicity or ototoxicity by virtue of limited absorption from the tissue bed. There is one retrospective study in the vascular surgery literature of 454 patients undergoing aortofemoral or infrainguinal procedures that showed reduction of 30-day SSI rates with use of topical vancomycin compared to controls (25.1 vs. 17.2%, p=0.049). More extensive data regarding the use of topical vancomycin prophylaxis comes from the orthopaedic literature. A recent review of orthopaedic studies, although mostly retrospective, highlighted benefits in spine surgery, total joint arthroplasty, foot and ankle surgery and elbow surgery. Further, 8 spine meta-analyses since 2014 have shown reduction in SSI rates with topical vancomycin administration.

Local gentamicin applied to surgical wounds has also been found effective, particularly in the prevention of gram-negative SSI, providing broad gram-negative coverage including Pseudomonas species. One randomized controlled trial assessing the prophylactic use of collagen gentamicin sponge in 40 patients undergoing prosthetic femoropopliteal bypass found significant reduction in groin SSI with use of a collagen gentamicin sponge (Collatamp G). An additional prospective cohort study and case series data also show favorable results in small patient samples of patients An additional prospective cohort study and case series data also show favorable results in small patient samples of patients undergoing various vascular operations. Cardiac surgeons have reported effective use of this antibiotic locally in prevention of sternal wound infections. Notably, a large randomized, double blinded-controlled trial of 1950 patients undergoing cardiac surgery through median sternotomy demonstrated decreased SSI rates at 60 days with the use of gentamicin containing collagen implants compared to controls (4.3 vs. 9.0%, p<0.001). The ability of gentamicin eluting sponges to prevent SSI in sternal wounds was confirmed in a recent meta-analysis. These sponges achieve high local levels of gentamicin for 36 hours with minimal systemic absorption in addition to accelerating hemostasis. Recently, wound closure using topical vancomycin paste and gentamicin irrigation has been shown in a retrospective study to reduce SSI in cardiac surgery sternotomy wounds by almost two thirds.

In this trial, an aggressive prophylactic approach using selective administration of topical vancomycin and gentamicin to the surgical wounds of patients undergoing open lower extremity revascularization at high-risk for SSI based on an elevated body mass index (BMI) >30, tissue loss, redo surgery, diabetes mellitus or renal failure will be compared to similar patients receiving standard perioperative antibiotic prophylaxis and wound care to evaluate the impact on 90-day SSI rates.

ELIGIBILITY:
Inclusion Criteria:

Patients identified as requiring lower extremity bypass for peripheral arterial disease by their consultant surgeon with high-risk features for vascular surgical site infection including,

* BMI >30
* Dialysis dependence
* Redo surgery
* Diabetes mellitus (type 1 or 2)
* Tissue loss (ischemic ulceration or gangrene of the feet)

Exclusion Criteria:

* Patient does not provide informed consent for surgery or study
* Patient received antibiotics for an active infection within 7 days prior to surgery
* Patient has an allergy to gentamicin or vancomycin
* Patient has a pre-existing infection of the surgical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with surgical site infection (%) | 90 days
  Per CDC definition and according to Szilagyi classification

SECONDARY OUTCOMES:
Length of stay | Perioperative period
  In-hospital following initial surgery
Number of Emergency Department Visits | 90 days
  Between discharge and first post-operative follow-up appointment
Number of participants dying of any cause | 90 days
  Any cause
Number of participants requiring re-operation | 90 days
  For graft failure
Number of participants requiring major lower limb amputation | 90 days
  Above ankle

CONTACTS AND LOCATIONS:
Overall Officials: Luc Dubois, MD, MSc, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen LL, Brahmanandam S, Bandyk DF, Belkin M, Clowes AW, Moneta GL, Conte MS. Female gender and oral anticoagulants are associated with wound complications in lower extremity vein bypass: an analysis of 1404 operations for critical limb ischemia. J Vasc Surg. 2007 Dec;46(6):1191-1197. doi: 10.1016/j.jvs.2007.07.053. PMID 18154995
- [Background] Giles KA, Hamdan AD, Pomposelli FB, Wyers MC, Siracuse JJ, Schermerhorn ML. Body mass index: surgical site infections and mortality after lower extremity bypass from the National Surgical Quality Improvement Program 2005-2007. Ann Vasc Surg. 2010 Jan;24(1):48-56. doi: 10.1016/j.avsg.2009.05.003. Epub 2009 Jul 19. PMID 19619975
- [Background] Greenblatt DY, Rajamanickam V, Mell MW. Predictors of surgical site infection after open lower extremity revascularization. J Vasc Surg. 2011 Aug;54(2):433-9. doi: 10.1016/j.jvs.2011.01.034. Epub 2011 Mar 31. PMID 21458203
- [Background] Vogel TR, Dombrovskiy VY, Carson JL, Haser PB, Lowry SF, Graham AM. Infectious complications after elective vascular surgical procedures. J Vasc Surg. 2010 Jan;51(1):122-9; discussion 129-30. doi: 10.1016/j.jvs.2009.08.006. Epub 2009 Dec 2. PMID 19954920
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Background] Turtiainen J, Hakala T. Surgical wound infections after peripheral vascular surgery. Scand J Surg. 2014 Dec;103(4):226-31. doi: 10.1177/1457496913514384. Epub 2014 Apr 15. PMID 24737857
- [Background] Bandyk DF. Vascular surgical site infection: risk factors and preventive measures. Semin Vasc Surg. 2008 Sep;21(3):119-23. doi: 10.1053/j.semvascsurg.2008.05.008. PMID 18774446
- [Background] Pevzner L, Swank M, Krepel C, Wing DA, Chan K, Edmiston CE Jr. Effects of maternal obesity on tissue concentrations of prophylactic cefazolin during cesarean delivery. Obstet Gynecol. 2011 Apr;117(4):877-882. doi: 10.1097/AOG.0b013e31820b95e4. PMID 21422859
- [Background] Ott E, Bange FC, Sohr D, Teebken O, Mattner F. Risk factors associated with surgical site infections following vascular surgery at a German university hospital. Epidemiol Infect. 2013 Jun;141(6):1207-13. doi: 10.1017/S095026881200180X. Epub 2012 Aug 21. PMID 22906362
- [Background] Siracuse JJ, Nandivada P, Giles KA, Hamdan AD, Wyers MC, Chaikof EL, Pomposelli FB, Schermerhorn ML. Prosthetic graft infections involving the femoral artery. J Vasc Surg. 2013 Mar;57(3):700-5. doi: 10.1016/j.jvs.2012.09.049. Epub 2013 Jan 9. PMID 23312940
- [Background] Virkkunen J, Heikkinen M, Lepantalo M, Metsanoja R, Salenius JP; Finnvasc Study Group. Diabetes as an independent risk factor for early postoperative complications in critical limb ischemia. J Vasc Surg. 2004 Oct;40(4):761-7. doi: 10.1016/j.jvs.2004.07.040. PMID 15472606
- [Background] Ramdev P, Rayan SS, Sheahan M, Hamdan AD, Logerfo FW, Akbari CM, Campbell DR, Pomposelli FB Jr. A decade experience with infrainguinal revascularization in a dialysis-dependent patient population. J Vasc Surg. 2002 Nov;36(5):969-74. doi: 10.1067/mva.2002.128297. PMID 12422107
- [Background] Khan NR, Thompson CJ, DeCuypere M, Angotti JM, Kalobwe E, Muhlbauer MS, Camillo FX, Klimo P Jr. A meta-analysis of spinal surgical site infection and vancomycin powder. J Neurosurg Spine. 2014 Dec;21(6):974-83. doi: 10.3171/2014.8.SPINE1445. Epub 2014 Sep 26. PMID 25259555
- [Background] Mohammed S, Pisimisis GT, Daram SP, Bechara CF, Barshes NR, Lin PH, Kougias P. Impact of intraoperative administration of local vancomycin on inguinal wound complications. J Vasc Surg. 2013 Apr;57(4):1079-83. doi: 10.1016/j.jvs.2012.09.073. Epub 2013 Jan 11. PMID 23313181
- [Background] Fleischman AN, Austin MS. Local Intra-wound Administration of Powdered Antibiotics in Orthopaedic Surgery. J Bone Jt Infect. 2017 Jan 1;2(1):23-28. doi: 10.7150/jbji.16649. eCollection 2017. PMID 28529861
- [Background] Ghobrial GM, Cadotte DW, Williams K Jr, Fehlings MG, Harrop JS. Complications from the use of intrawound vancomycin in lumbar spinal surgery: a systematic review. Neurosurg Focus. 2015 Oct;39(4):E11. doi: 10.3171/2015.7.FOCUS15258. PMID 26424335
- [Background] Alcala-Cerra G, Paternina-Caicedo AJ, Moscote-Salazar LR, Gutierrez-Paternina JJ, Nino-Hernandez LM. [Application of vancomycin powder into the wound during spine surgery: systematic review and meta-analysis]. Rev Esp Cir Ortop Traumatol. 2014 May-Jun;58(3):182-91. doi: 10.1016/j.recot.2013.10.004. Epub 2014 Apr 2. Spanish. PMID 24703108
- [Background] Xiong L, Pan Q, Jin G, Xu Y, Hirche C. Topical intrawound application of vancomycin powder in addition to intravenous administration of antibiotics: A meta-analysis on the deep infection after spinal surgeries. Orthop Traumatol Surg Res. 2014 Nov;100(7):785-9. doi: 10.1016/j.otsr.2014.05.022. Epub 2014 Oct 3. PMID 25281550
- [Background] Kang DG, Holekamp TF, Wagner SC, Lehman RA Jr. Intrasite vancomycin powder for the prevention of surgical site infection in spine surgery: a systematic literature review. Spine J. 2015 Apr 1;15(4):762-70. doi: 10.1016/j.spinee.2015.01.030. Epub 2015 Jan 28. PMID 25637469
- [Background] Chiang HY, Herwaldt LA, Blevins AE, Cho E, Schweizer ML. Effectiveness of local vancomycin powder to decrease surgical site infections: a meta-analysis. Spine J. 2014 Mar 1;14(3):397-407. doi: 10.1016/j.spinee.2013.10.012. Epub 2013 Oct 30. PMID 24373682
- [Background] Bakhsheshian J, Dahdaleh NS, Lam SK, Savage JW, Smith ZA. The use of vancomycin powder in modern spine surgery: systematic review and meta-analysis of the clinical evidence. World Neurosurg. 2015 May;83(5):816-23. doi: 10.1016/j.wneu.2014.12.033. Epub 2014 Dec 19. PMID 25535069
- [Background] Evaniew N, Khan M, Drew B, Peterson D, Bhandari M, Ghert M. Intrawound vancomycin to prevent infections after spine surgery: a systematic review and meta-analysis. Eur Spine J. 2015 Mar;24(3):533-42. doi: 10.1007/s00586-014-3357-0. Epub 2014 May 18. PMID 24838506
- [Background] Hussain ST. Local application of gentamicin-containing collagen implant in the prophylaxis and treatment of surgical site infection following vascular surgery. Int J Surg. 2012;10 Suppl 1:S5-9. doi: 10.1016/j.ijsu.2012.05.015. Epub 2012 May 29. PMID 22659222
- [Background] Horch R, Kronung G. [Prevention of infection in teflon prostheses for dialysis access. Experiences with a resorbable combined collagen-antibiotic system]. Vasa. 1989;18(1):30-4. German. PMID 2929171
- [Background] Holdsworth J. Treatment of infective and potentially infective complications of vascular bypass grafting using gentamicin with collagen sponge. Ann R Coll Surg Engl. 1999 May;81(3):166-70. PMID 10364947
- [Background] Friberg O, Svedjeholm R, Soderquist B, Granfeldt H, Vikerfors T, Kallman J. Local gentamicin reduces sternal wound infections after cardiac surgery: a randomized controlled trial. Ann Thorac Surg. 2005 Jan;79(1):153-61; discussion 161-2. doi: 10.1016/j.athoracsur.2004.06.043. PMID 15620935
- [Background] Kowalewski M, Pawliszak W, Zaborowska K, Navarese EP, Szwed KA, Kowalkowska ME, Kowalewski J, Borkowska A, Anisimowicz L. Gentamicin-collagen sponge reduces the risk of sternal wound infections after heart surgery: Meta-analysis. J Thorac Cardiovasc Surg. 2015 Jun;149(6):1631-40.e1-6. doi: 10.1016/j.jtcvs.2015.01.034. Epub 2015 Jan 23. PMID 25703409
- [Background] Ruszczak Z, Friess W. Collagen as a carrier for on-site delivery of antibacterial drugs. Adv Drug Deliv Rev. 2003 Nov 28;55(12):1679-98. doi: 10.1016/j.addr.2003.08.007. PMID 14623407
- [Background] Andreas M, Muckenhuber M, Hutschala D, Kocher A, Thalhammer F, Vogt P, Fleck T, Laufer G. Direct sternal administration of Vancomycin and Gentamicin during closure prevents wound infection. Interact Cardiovasc Thorac Surg. 2017 Jul 1;25(1):6-11. doi: 10.1093/icvts/ivx032. PMID 28402472
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835